CLINICAL TRIAL: NCT05643495
Title: A Phase 2, Open-label Study Evaluating Efficacy and Safety of VX-864 in Subjects With Alpha-1 Antitrypsin Deficiency Who Have the PiZZ Genotype, Over 48 Weeks
Brief Title: A Study to Evaluate Efficacy and Safety of VX-864 in Participants With the PiZZ Genotype
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study drug dosing was permanently discontinued at the Sponsor's discretion based on frequency and nature of skin and subcutaneous tissue disorders.
Sponsor: Vertex Pharmaceuticals Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: VX22-864-108; 2022-002746-40 (EudraCT Number)
Record Dates: First submitted 2022-11-29; First posted 2022-12-08 (Actual); Results first posted 2025-09-08 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-08

CONDITIONS: Alpha-1 Antitrypsin Deficiency
MeSH Terms: conditions — alpha 1-Antitrypsin Deficiency

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): Participants received VX-864 every 12 hours (q12h) for 48 weeks or until study drug dosing was terminated.
  Interventions: Drug: VX-864
- Group B (Experimental): Participants undergo a liver biopsy before receiving VX-864 q12h for 48 weeks or until study drug dosing was terminated, and undergo a second liver biopsy at either Week 24 or Week 48.
  Interventions: Drug: VX-864

INTERVENTIONS:
Drug: VX-864 — Tablets for oral administration.

SUMMARY:
The purpose of this study evaluates the efficacy and safety of VX-864 in participants with the PiZZ genotype over 48 weeks.

ELIGIBILITY:
Key Inclusion Criteria:

* Participants must have a PiZZ genotype confirmed at screening
* Plasma AAT levels indicating severe deficiency at screening

Key Exclusion Criteria:

* History of a medical condition that could negatively impact the ability to complete the study
* Solid organ, or hematological transplantation or is currently on a transplant list
* History of use of gene therapy or Ribonucleic acid interference (RNAi) therapy at any time previously
* Participants for whom discontinuation of augmentation therapy is not considered to be in their best interest, based on the clinical judgement of the treating physician

Other protocol defined Inclusion/Exclusion criteria may apply.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2023-02-23 (Actual); Primary Completion 2024-08-19 (Actual); Study Completion 2024-08-19 (Actual)

CONTACTS AND LOCATIONS:
Locations (13):
- United States (10):
  - University of Florida, Gainesville, Florida
  - Central Florida Pulmonary Group, P.A., Orlando, Florida
  - The University of Iowa Hospitals and Clinics: Adult Pulmonary Clinic, Iowa City, Iowa
  - University of Kansas Medical Center, Kansas City, Kansas
  - Hannibal Regional Healthcare System, Hannibal, Missouri
  - Columbia University Irving Medical Center, New York, New York
  - Marsico Clinical Research Center at UNC Pulmonary Clinic, Chapel Hill, North Carolina
  - Renovatio Clinical, Houston, Texas
  - University of Utah Health, Salt Lake City, Utah
  - Inova Fairfax Medical Campus, Falls Church, Virginia
- University Hospital RWTH Aachen, Aachen, Germany
- Royal College of Surgeons in Ireland Clinical Research Centre, Beaumont Hospital, Beaumont, Ireland
- King's College Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Details on Vertex data sharing criteria and process for requesting access can be found at: https://www.vrtx.com/independent-research/clinical-trial-data-sharing

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study had 2 Groups: Group A participants did not have a liver biopsy and Group B participants have 2 liver biopsies performed over the course of the study.
Pre-assignment Details: A total of 14 participants were enrolled from 23 February 2023 to 03 November 2023 in this study. Study drug dosing and efficacy assessments were terminated early due to Sponsor decision, therefore evaluation of efficacy outcome measure was not completed.
Groups:
- Group A VX-864 500 mg: Participants received VX-864 every 12 hours (q12h) for 48 weeks or until study drug dosing was terminated.
- Group B VX-864 500 mg: Participants undergo a liver biopsy before receiving VX-864 q12h for 48 weeks or until study drug dosing was terminated and undergo a second liver biopsy at either Week 24 or Week 48.
Period: Overall Study
Arm/Group | Group A VX-864 500 mg | Group B VX-864 500 mg
Started | 10 | 4
Completed | 9 | 2
Not Completed | 1 | 2
Not completed — Adverse Event | 0 | 1
Not completed — Withdrawal of consent (not due to AE) | 1 | 1

BASELINE CHARACTERISTICS:
Population: The Full Analysis Set (FAS) is defined as all enrolled participants who have received at least 1 dose of study drug.
Groups:
- Group A VX-864 500 mg: Participants received VX-864 q12h for 48 weeks or until study drug dosing was terminated.
- Total: Total of all reporting groups
Arm/Group | Group A VX-864 500 mg | Group B VX-864 500 mg | Total
Number analyzed (Participants) | 10 | 4 | 14
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.8 (14.2) | 50.8 (10.4) | 52.2 (12.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 3 | 11
  Male | 2 | 1 | 3
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 10 | 4 | 14
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Not Hispanic or Latino | 10 | 4 | 14

OUTCOME MEASURES:

1. Primary Outcome: Change in Blood Functional Alpha-1 Antitrypsin (AAT) Levels
Time Frame: From Baseline at Week 48
Population: Data was not collected for this Outcome Measure as the study drug dosing was terminated prior to any participant reaching Week 48.
Arm/Group | Group A VX-864 500 mg | Group B VX-864 500 mg
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Change in Blood Functional AAT Levels
Time Frame: From Baseline up to Week 48
Population: as for outcome 1
Arm/Group | Group A VX-864 500 mg | Group B VX-864 500 mg
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Change in Blood Antigenic AAT Levels
Time Frame: From Baseline up to Week 48
Population: as for outcome 1
Arm/Group | Group A VX-864 500 mg | Group B VX-864 500 mg
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Change in Blood Z-polymer Levels
Time Frame: From Baseline up to Week 48
Population: as for outcome 1
Arm/Group | Group A VX-864 500 mg | Group B VX-864 500 mg
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Group B: Change in Z-polymer Accumulation in the Liver
Time Frame: From Baseline up to Week 48
Population: No participants in Group B underwent a second liver biopsy at week 24 or week 48 as the study drug dosing was terminated prior to any participant reaching week 24 or week 48. Therefore, data was not collected for this Outcome Measure.
Arm/Group | Group A VX-864 500 mg | Group B VX-864 500 mg
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Safety and Tolerability as Assessed by Number of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs)
Time Frame: Day 1 up to Week 52
Population: Safety set included all participants who had received at least 1 dose of study drug in this study.
Measure: Count of Participants; unit: Participants
Arm/Group | Group A VX-864 500 mg | Group B VX-864 500 mg
Number analyzed (Participants) | 10 | 4
Participants
  Participants with TEAEs | 10 | 4
  Participants with SAEs | 1 | 0

ADVERSE EVENTS:
Time Frame: Day 1 up to Week 52
Description: Safety set included all participants who had received at least 1 dose of study drug in this study.
Arm/Group | Group A VX-864 500 mg | Group B VX-864 500 mg
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/4
Serious Adverse Events (participants affected / at risk) | 1/10 | 0/4
Other Adverse Events (participants affected / at risk) | 10/10 | 4/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Group A VX-864 500 mg (N=10) | Group B VX-864 500 mg (N=4)
Diverticulitis (Infections and infestations) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Group A VX-864 500 mg (N=10) | Group B VX-864 500 mg (N=4)
Porphyria non-acute (Congenital, familial and genetic disorders) | 0 | 1
Abdominal distension (Gastrointestinal disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 2 | 2
Mouth ulceration (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 3 | 2
Paraesthesia oral (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 1
Hypertransaminasaemia (Hepatobiliary disorders) | 1 | 0
Bronchitis (Infections and infestations) | 0 | 1
Diverticulitis (Infections and infestations) | 1 | 0
Blood creatine phosphokinase increased (Investigations) | 1 | 1
Hypercholesterolaemia (Metabolism and nutrition disorders) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 1
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 | 0
Dizziness (Nervous system disorders) | 2 | 0
Dysgeusia (Nervous system disorders) | 1 | 0
Headache (Nervous system disorders) | 0 | 1
Hyperaesthesia (Nervous system disorders) | 1 | 0
Irritability (Psychiatric disorders) | 1 | 0
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1 | 0
Blister (Skin and subcutaneous tissue disorders) | 2 | 0
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 | 0
Drug eruption (Skin and subcutaneous tissue disorders) | 1 | 0
Dyshidrotic eczema (Skin and subcutaneous tissue disorders) | 1 | 0
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 3 | 0
Post inflammatory pigmentation change (Skin and subcutaneous tissue disorders) | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0
Pseudoporphyria (Skin and subcutaneous tissue disorders) | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 1
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2023-11-02): https://cdn.clinicaltrials.gov/large-docs/95/NCT05643495/Prot_000.pdf
  • Statistical Analysis Plan (2023-11-30): https://cdn.clinicaltrials.gov/large-docs/95/NCT05643495/SAP_001.pdf